CLINICAL TRIAL: NCT03252717
Title: Radiation-induced Late Side-effects: Predictive Role of New Biomarkers for Selecting Hypersensitive Patients to Ionizing Radiation in Breast Cancer (BIORISE)
Brief Title: Predictive Role of New Biomarkers for Hypersensitive Patients to Radiation in Breast Cancer (BIORISE)
Acronym: BIORISE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICM-URC-2014/22
Record Dates: First submitted 2016-08-29; First posted 2017-08-17 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- blood sample (Experimental): Pre-treatment blood samples will be collected: 8 samples
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Pre-treatment blood samples will be collected for downstream analyses:
  * Three 6 ml EDTA samples for proteomic and genomic work package
  * One 6 ml dry sample for auto-antibodies analysis in the immunology work package
  * Two 4 ml EDTA samples for DNA extraction in the immunology work package
  * Two 2.5 ml PAX Gene sample for RNA extraction in the immunology work package and the non-irradiated control in the genomic work package

SUMMARY:
To confirm the protein expression level in radiation-induced late effects patients and to determine the performance value, in particular the positive predictive value, of a blood test based on the dosage of a panel of five proteins, it is necessary to validate these preliminary results by a prospective study on a large cohort of patients.

DETAILED DESCRIPTION:
Molecular mechanisms involved in radiation-induced responses are complex, and proteomic approaches can be used to better understand the overall reaction process of ionizing radiation and to identify potential radio-sensitive predictive markers. Until now, few publications have addressed the determination of radiosensitive patients.

Based on our previous results and in order to improve the positive predictive value of the radiation induced late effect assay, we developed a quantitative proteomic approach to identify predictive radiobiological markers in patients with severe toxicity. First, four patients were selected with a low RILA value from the prospective studies mentioned above. Two patients had no toxicity at least four years after the end of treatment whereas two others patients developed a severe toxicity greater than grade 2. T-lymphocytes have been isolated from whole blood and half of them have been irradiated in vitro. It will then performed a quantitative proteomics workflow using an 8-plex iTRAQ labeling and after several fractionations to optimize resolution of analysis (off gel fractionation followed by nanoliquid chromatography), proteins were identified by tandem mass spectrometry (4800 plus MALDI TOF/TOF). More than 1300 total proteins were identified with high confidence (95%, one unique peptide). At 0 Gy, 135 proteins were differentially expressed between patients with or without severe radio-induced toxicity. In irradiated T-lymphocytes (8 Gy), 107 proteins were differentially expressed between patients with or without severe radio-induced toxicity. Among them, five proteins (AK2, adenylate kinase 2; IDH2, isocitrate dehydrogenase 2 (NADP+); ANX1, annexin 1; APEX1, DNA-(apurinic or apyrimidinic site) lyase, and HSC70, Heat shock cognate 71 kDa) with the highest protein expression ratio (>1.5) and that showed no difference expression ratio in 0 Gy controls, were selected for consecutive validation. These proteins are involved in several mechanisms including metabolism and energy production, apoptosis, calcium binding protein, and DNA damages repair. These five proteins are currently the subject of patent application.

Then,10 other patients will be recruited (5 patients with grade ≥ 2 breast fibrosis and 5 patients without toxicity) who presented a low RILA value to validate proteins expression by western-blotting. Results showed that all proteins were overexpressed in irradiated T-lymphocytes patients with severe toxicity comparatively to patients without toxicity.

However, to confirm the protein expression level in radiation-induced late effects patients and to determine the performance value, in particular the positive predictive value, of a blood test based on the dosage of a panel of five proteins, it is necessary to validate these preliminary results by a prospective study on a large cohort of patients

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for adjuvant radiotherapy for cancer of the breast (invasive or in situ) including breast patients receiving neo-adjuvant chemotherapy. Patients receiving chemotherapy should have completed their course of chemotherapy (anthracyclines) at least one month prior to radiotherapy commencing.
* No other malignancy prior to treatment for the specified tumour types except basal cell or squamous cell carcinoma of the skin
* No evidence of distant metastases
* Patients able to provide a venous blood sample
* Willingness and ability to comply with scheduled visits, treatment plans and available for follow up
* Greater than 18 years of age; no upper age limit
* The capacity to understand the patient information sheet and the ability to provide written informed consent
* Patients must be affiliated to a Social Security System

Exclusion Criteria:

* Patients with metastatic disease
* Prior irradiation at the same site
* Planned use of protons
* Breast patients receiving concomitant chemo-radiation
* Male breast cancer patients
* Mastectomy patients
* Bilateral breast cancer
* Mental disability or patient otherwise unable to give informed consent
* Limited life expectancy due to co-morbidity
* Pregnant patients
* Partial breast irradiation
* Patients with breast implants if not removed during surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
blood sample to assess dosage of 5 proteins | through study completion, an average of 5 years
  Confirm the predictive value, of a blood test based on the dosage of a panel of five (5) proteins: AK2 - IDH2 - ANX1- APEX1 - HSC70 in radiation-induced late side effects after breast-conserving surgery and curative intent adjuvant radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: david azria, Study Chair — Institut régional du Cancer de Montpellier
Locations (1):
- Institut régional du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No